CLINICAL TRIAL: NCT03576404
Title: The Impact of Comprehensive Medication Review by Pharmacist in Hemodialysis Patients: A Quasi Experimental Interrupted Time Series Study
Brief Title: Patient-Centered Pharmacist Care in the Hemodialysis Unit: A Quasi-Experimental Interrupted Time Series Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: Harvard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SP16/099/J
Record Dates: First submitted 2018-04-26; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-04

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: A Quasi-Experimental Interrupted Time Series Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible participants (Experimental): The intervention of patient-centered pharmacist care included a comprehensive interview patients conducted at month 3 and 5 ,which included and reviewing all their medications using concepts of MTM and MI All study participants were assessed at baseline and on monthly basis for the changes in the study outcomes.
  Interventions: Other: Patient-Centered Pharmacist Care

INTERVENTIONS:
Other: Patient-Centered Pharmacist Care — A comprehensive interview applying the concepts of Medication Therapy Management (MTM) and Motivational Interview (MI)

SUMMARY:
Nonadherence to medications by patients requiring hemodialysis (HD) leads to unfavorable clinical outcomes.Limited data exist on the influence of pharmacists on pharmacoadherence by patients requiring HD. Therefore, we assessed the impact of patient-centered pharmacist care through the implementation of concepts of Medication Therapy Management (MTM) and motivational interview (MI) on pharmacoadherence and its outcomes in patients requiring HD.

DETAILED DESCRIPTION:
Patients were assessed at baseline for baseline characteristics, dialysis-related factors, and medications records

1. Pharmacists conducted brief monthly interview for patients to assess the medications they are receiving
2. A comprehensive interview for patients occurred at month 3 and 5 including concepts of MTM and MI
3. MTM included a review of each participant's medications and personal medication record to identify the use of any over-the-counter medications, design of their medication-related action plan, formulation of specific therapeutic interventions, and referrals for discussion with their physician and subsequent documentation and follow-up. The therapeutic interventions accepted by the physician were further discussed with each patient/caregiver using the MI technique to encourage adherence and this discussion was documented in each patient's medication record.
4. MI incorporated the main components reported in the literature: rolling with resistance; expressing empathy; avoiding argumentative behavior; highlighting the discrepancy between patients' current attitudes compared with the desired therapeutic goals; and empowering patients' self-efficacy

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥18 years of age)
* Outpatient HD for at least 3 months before the study period

Exclusion Criteria:

* Patients who refused to participate in the study
* Patients without the capacity to understand or take responsibility for their medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-04-23 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in pharmacoadherence of patients requiring HD using electronic medication refill from baseline | Monthly and up to 6 months
  Comparing changes in self-reporting of number of medications with electronic prescribing during each of the six interviews
Changes in pharmacoadherence of patients requiring HD through the control of serum phosphate level (mmol/L) from baseline | Monthly and up to 6 months
  Changes in surrogate laboratory pre-HD serum phosphate level (mmol/L) from baseline

SECONDARY OUTCOMES:
Changes in Systolic blood pressure (SBP) control in mmHg from baseline as a independent surrogate marker for administration of medications | Monthly and up to 6 months
  Changes in Systolic blood pressure (SBP) control in mmHg from baseline and on a monthly basis
Changes in serum low-density lipoprotein (LDL) levels in mmol/L from baseline as an independent surrogate marker for the administration of medications | Monthly and up to 6 months
  Changes in serum low-density lipoprotein (LDL) levels in mmol/L from baseline and on a monthly basis
Changes in Number of Medication-related problems (MRPs) from baseline at month 3 and month 5 | At month 3 and month 5 of the study
  Number
Types of Medication-related problems (MRPs) | Total study duration: from month 1 to month 6
  Types of Medication-related problems included in the study as identified in literature: improper drug dosing or selection; initiation of medication without indication; adverse drug events; failure to receive drugs; indication without treatment; suggested alternative therapeutic options; and inappropriate monitoring or laboratory tests required
Number of accepted therapeutic interventions by the pharmacist | Monthly and up to 6 months
  Number of Therapeutic interventions suggested by the pharmacists to alter medication regimen suggested by pharmacist based on discussion and approval of prescribing physicians

CONTACTS AND LOCATIONS:
Overall Officials: Sherine E Ismail, PharmD, MPH, Principal Investigator — KAIMRC, King Saud bin Abdulaziz University for Health Sciences, Pharmaceutical Care Department, King Khalid Hospital, Ministry of National Guard Health Affairs, Jeddah, Saudi Arabia, Harvard T. H. Chan School of Public Health, Boston, MA, USA

IPD SHARING:
Plan to Share IPD: Yes
I plan to share the listed below data regarding my study for public upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication, I can share all the supporting information
Access Criteria: After publication

REFERENCES:
- [Derived] Ismail S, Al-Subhi A, Youssif E, Ahmed M, Almalki A, Seger DL, Seger AC, Cook E. Patient-centered Pharmacist Care in the Hemodialysis Unit: a quasi-experimental interrupted time series study. BMC Nephrol. 2019 Nov 13;20(1):408. doi: 10.1186/s12882-019-1577-6. PMID 31722680